CLINICAL TRIAL: NCT00164398
Title: HIP: HIV Intervention for Providers
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: CDC-NCHSTP-3986; CCR 920974
Record Dates: First submitted 2005-09-09; First posted 2005-09-14 (Estimated); Last update posted 2012-09-11 (Estimated); Status verified 2012-09

CONDITIONS: HIV Infections
Keywords: HIV
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: HIP: HIV Intervention for Providers

SUMMARY:
The purpose is to encourage Provider participants to evaluate high risk HIV transmission behaviors and offer prevention messages to their HIV+ patients which will, in turn, reduce rates of unprotected anal and/or vaginal sex with partners of known HIV sero-negativity or unknown HIV serostatus. It is hypothesized that patients of providers participating in the HIP intervention will report higher reduction in sexual risk practices, when compared to the patients of the providers who were randomized into the control condition.

ELIGIBILITY:
Inclusion Criteria:

* Provider participants: (1) licensed MD, NP or PA on staff at the participating institution; (2) has a minimum panel of 5 HIV+ patients; (3) sees patients at least one-half day per week in the clinical setting; (4) is willing to participate in all intervention training sessions; and (5) is willing and able to provide full informed consent.

HIV+ patient participants:(1) report at least 1 encounter of unprotected anal or vaginal sex with known HIV- or unknown serostatus partner in the preceding six months; (2) patient's Primary Provider is enrolled as a participant in the study; (3) age 18 years or older; and (4) willing and able to provide informed consent.

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2004-06; Primary Completion 2006-10 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
Self-reported, unprotected (without condoms) anal or vaginal sex with HIV-negative and unknown-status persons.

CONTACTS AND LOCATIONS:
Overall Officials: Dogan Eroglu, PhD., Principal Investigator — Centers for Disease Control and Prevention
Locations (1):
- University of California San Francisco - CAPS, San Francisco, California, United States

REFERENCES:
- [Derived] Rose CD, Courtenay-Quirk C, Knight K, Shade SB, Vittinghoff E, Gomez C, Lum PJ, Bacon O, Colfax G. HIV intervention for providers study: a randomized controlled trial of a clinician-delivered HIV risk-reduction intervention for HIV-positive people. J Acquir Immune Defic Syndr. 2010 Dec 15;55(5):572-81. doi: 10.1097/QAI.0b013e3181ee4c62. PMID 20827218